CLINICAL TRIAL: NCT01764256
Title: A Phase 1 Double Blinded, Randomized, Placebo-controlled Dose Escalation Study to Examine the Safety, Reactogenicity, Tolerability and Immunogenicity of the P2-VP8 Subunit Rotavirus Vaccine in Healthy Adult Volunteers
Brief Title: A Phase 1 Dose Escalation Study to Examine the Safety of the P2-VP8 Rotavirus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC 009
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Rotavirus Infection
Keywords: rotavirus; vaccine
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 10 μg P2-VP8 (Experimental): 3 doses of P2-VP8 subunit rotavirus vaccine (Lot # 1746) produced in E. coli was adsorbed onto aluminum hydroxide (0.6 mg/dose) adjuvant prior to administration. Each dose contained 10 μg of active ingredient.
  Interventions: Biological: P2-VP8 subunit rotavirus vaccine
- 30 μg P2-VP8 (Experimental): 3 doses of P2-VP8 subunit rotavirus vaccine (Lot # 1746) produced in E. coli was adsorbed onto aluminum hydroxide (0.6 mg/dose) adjuvant prior to administration. Each dose contained 30 μg of active ingredient.
  Interventions: Biological: P2-VP8 subunit rotavirus vaccine
- 60 μg P2-VP8 (Experimental): 3 doses of P2-VP8 subunit rotavirus vaccine (Lot # 1746) produced in E. coli was adsorbed onto aluminum hydroxide (0.6 mg/dose) adjuvant prior to administration. Each dose contained 60 μg of active ingredient.
  Interventions: Biological: P2-VP8 subunit rotavirus vaccine
- Placebo (Placebo Comparator): 3 doses of placebo delivered intramuscularly.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: P2-VP8 subunit rotavirus vaccine — P2-VP8 subunit rotavirus vaccine was made by inserting a codon optimized synthetic gene for the VP8 region of rotavirus VP4 fused to the P2 T-cell epitope of tetanus toxin into the Pj411 proprietary cloning vector developed by DNA 2.0, Menlo Park, CA. The vector carries a kanamycin resistance gene as a selection marker. The vector was transfected into the BL21 strain of E. coli. The fusion protein was purified from Isopropyl β-D-1-thiogalactopyranoside (IPTG)-induced and physically lysed cultures using standard column chromatographic techniques employing Q-Sepharose and Butyl 650 as resins in addition to ultrafiltration and diafiltration.
  Arms: 10 μg P2-VP8; 30 μg P2-VP8; 60 μg P2-VP8
Other: placebo — Sodium Chloride 0.9%, USP for Injection was used to dilute the active P2-VP8 vaccine to final dosing concentration and was used for the Placebo for the study.
  Arms: Placebo

SUMMARY:
This study will evaluate 3 doses of a new vaccine for rotavirus infection in healthy adult volunteers to determine if it is safe and if the immune systems of healthy adults respond to this vaccine.

DETAILED DESCRIPTION:
The trial will be a double-blinded, randomized, placebo-controlled dose-escalation study in which three dose-levels of vaccine will be tested in adults. Cohorts of 16 individuals (12 vaccine recipients and 4 placebo recipients) per dose level will receive three intramuscular injections four weeks apart. The three dose levels of vaccine to test will be 10 microgram (μg), 30 μg and 60 μg.

ELIGIBILITY:
Inclusion Criteria:

* A qualified volunteer must be:

  1. Healthy male or female between 18 and 45 (inclusive) years of age at time of enrollment.
  2. Willing and able to give informed consent - must pass test of comprehension with > 70% correct within two attempts.
  3. If female and of childbearing potential, be not breastfeeding and not pregnant (based on a negative serum pregnancy test at screening and a negative urine pregnancy test during the 24 hours prior to first injection), planning to avoid pregnancy for at least 4 weeks after the last injection, and willing to use an adequate method of contraception consistently and have repeated pregnancy tests prior to second and third injections.
  4. Willing to comply with study restrictions and study schedule (as evidenced by a signed informed consent form (ICF) and assessment by the Principal Investigator (PI) or designee).
  5. Able and willing to be contacted by telephone or text, and willing for study staff to record telephone voice or text messages as needed.

     Exclusion Criteria:
* A qualified volunteer must not:

  1. Have received an investigational product during the 30 days prior to randomization.
  2. Intend to receive another investigational product during this study.
  3. Have any contraindication to parenteral injections (e.g., history of bleeding disorder).
  4. Have previously received a marketed or investigational rotavirus vaccine.
  5. Have a history of severe local or systemic reaction to any vaccine.
  6. Have a history of recurrent urticaria of unknown cause.
  7. Have a history of any allergic or infusion reaction that was severe (e.g., anaphylactic or anaphylactoid), generalized (e.g., drug rash, urticaria, angioedema) or that, in the opinion of the PI, significantly increases risk of severe local or systemic reaction to an investigative vaccine.
  8. Have a history of reaction to any vaccine that, in the opinion of the PI, significantly increases risk of severe reaction to an investigative vaccine.
  9. Have received any vaccine within 4 weeks prior to randomization or planned vaccination through Day 84.
  10. Have received any blood product or any immunomodulating agent (e.g., immunoglobulin, interferon, growth factor) within 12 weeks prior to randomization.
  11. Have received immunosuppressive medications (e.g., prolonged use of systemic corticosteroid or cytotoxic agent) within the 24 weeks prior to randomization. Eligible if a short course (≤10 days) of systemic corticosteroid concluded more than 2 weeks prior to randomization, use of inhaled corticosteroid for asthma, and use of topical corticosteroid for a skin condition.
  12. Have a history of any clinically significant (in the opinion of the PI) immunosuppressive or autoimmune condition.
  13. Anticipate need for administration of any blood product, immunosuppressive (e.g., systemic corticosteroid), or immunomodulatory treatment during the study.
  14. Have a history of malignancy, excluding basal cell carcinoma.
  15. Have Diabetes Mellitus Type I or II.
  16. Have a positive test for human immunodeficiency virus 1 (HIV-1), Hepatitis B surface antigen (HBsAg) or (Hepatitis C Antibody Test) anti-HepC.
  17. Have significant abnormalities in screening laboratory test results or clinical assessment as determined by the PI or by the PI in consultation with the Sponsor's medical officer.*
  18. Have abnormal vital signs deemed clinically relevant by the Principle Investigator (PI).
  19. Evidence of current or recent (within past 12 months) excessive alcohol consumption or drug dependence.
  20. Have any condition of hand, arm or related lymph nodes that may confound post-dose assessments.
  21. Have any condition (medical, psychiatric or behavioral) that, in the opinion of the PI, would increase the volunteer's health risks in study participation or would increase the risk of not achieving the study's objectives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Harro, MD, Principal Investigator — Johns Hopkins Bloomberg School of Hygiene and Public Health
Locations (1):
- Center for Immunization Research, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Fix AD, Harro C, McNeal M, Dally L, Flores J, Robertson G, Boslego JW, Cryz S. Safety and immunogenicity of a parenterally administered rotavirus VP8 subunit vaccine in healthy adults. Vaccine. 2015 Jul 17;33(31):3766-72. doi: 10.1016/j.vaccine.2015.05.024. Epub 2015 Jun 8. PMID 26065919

RESULTS

PARTICIPANT FLOW:
Period: Received All Vaccinations
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Started | 12 | 12 | 12 | 12
Completed | 10 | 11 | 11 | 12
Not Completed | 2 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Did not meet inclusion criteria | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Completed Study
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Started | 10 | 11 | 11 | 12
Completed | 10 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8 | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Full Range); unit: years] | 29.6 [19 to 39] | 34.2 [20 to 44] | 33.8 [24 to 42] | 32.5 [22 to 43] | 32.5 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 6 | 7 | 25
  Male | 5 | 7 | 6 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 48
Height [Mean (Full Range); unit: centimeters] | 172.7 [159 to 184] | 173.1 [157 to 189] | 168.8 [156 to 180] | 171.9 [160 to 188] | 171.6 [156 to 189]
Weight [Mean (Full Range); unit: kilograms] | 85.5 [49 to 135] | 90.0 [66 to 127] | 81.5 [57 to 101] | 85.6 [62 to 122] | 85.6 [49 to 135]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Severity of Adverse Events After Any Vaccination
Description: Adverse events were collected through 28 days following the final study injection and were graded for severity. Unsolicited adverse events were also assessed for relationship to vaccine. A final follow-up contact was attempted 6 months following the final study injection to inquire about new chronic health conditions, serious health events, and hospitalizations.
Time Frame: 6 months after final vaccination (224 days)
Measure: Count of Participants; unit: Participants
Arm/Group | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8 | Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Possibly related to vaccine: Mild | 1 | 2 | 0 | 2
  Possibly related to vaccine: Moderate | 0 | 1 | 0 | 0
  Possibly related to vaccine: Severe | 0 | 0 | 0 | 0
  Possibly related to vaccine: None | 11 | 9 | 12 | 10
  All adverse events: Mild | 6 | 2 | 6 | 5
  All adverse events: Moderate | 3 | 3 | 0 | 1
  All adverse events: Severe | 0 | 0 | 1 | 0
  All adverse events: None | 3 | 7 | 5 | 6
Statistical Analysis 1: Comparison: 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8 vs Placebo; Proportion of subjects with at least one unsolicited adverse event (related or unrelated); Test type: Equivalence — Definition of equivalence: p<0.05; p = 0.44, Fisher Exact
Statistical Analysis 2: Comparison: 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8 vs Placebo; Proportion of subjects with at least one unsolicited adverse event: potentially related; Test type: Equivalence — Definition of equivalence: p<0.05; p = 0.7446, Fisher Exact

2. Primary Outcome: Maximum Local or Systemic Reactogenicity After Any Vaccination
Description: For all cohorts, local and systemic reactogenicity data for all vaccinations were collected by subjects via diary card up to 7 days post each vaccination.
  Solicited systemic reactogenicity events included headache, muscle pain, fever, nausea, vomiting, fatigue, joint aches, and chills. Solicited local systemic reactogenicity events included injection site pain, tenderness, redness, swelling, itching, and local lymphadenopathy.
Time Frame: 7 days after each vaccination (Day 7, 35, 63)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  All reactogenicity: None | 7 | 3 | 6 | 4
  All reactogenicity: Mild | 3 | 7 | 6 | 6
  All reactogenicity: Moderate | 2 | 2 | 0 | 2
  Local reactogenicity: None | 7 | 4 | 7 | 4
  Local reactogenicity: Mild | 4 | 7 | 5 | 7
  Local reactogenicity: Moderate | 1 | 1 | 0 | 1
  Systemic reactogenicity: None | 10 | 4 | 9 | 6
  Systemic reactogenicity: Mild | 1 | 7 | 3 | 5
  Systemic reactogenicity: Moderate | 1 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic or local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 0.5694, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.0000, Fisher Exact

3. Primary Outcome: Maximum Local or Systemic Reactogenicity After the First Vaccination
Description: as for outcome 2
Time Frame: 7 days post Vaccination #1 on Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  All reactogenicity: None | 7 | 4 | 8 | 5
  All reactogenicity: Mild | 3 | 8 | 4 | 6
  All reactogenicity: Moderate | 2 | 0 | 0 | 1
  Local reactogenicity: None | 7 | 4 | 8 | 5
  Local reactogenicity: Mild | 4 | 8 | 4 | 6
  Local reactogenicity: Moderate | 1 | 0 | 0 | 1
  Systemic reactogenicity: None | 11 | 8 | 11 | 7
  Systemic reactogenicity: Mild | 0 | 4 | 1 | 5
  Systemic reactogenicity: Moderate | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic or local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 0.6004, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.00, Fisher Exact

4. Primary Outcome: Maximum Local or Systemic Reactogenicity After the Second Vaccination
Description: as for outcome 2
Time Frame: 7 days post Vaccination #2 on Day 35
Population: 47 subjects received the second vaccination (one less than Analysis Population Description). Subject in the placebo group withdrew Completed vaccination # 1 but withdrew due to moderate pain, tenderness and swelling, before Vaccination 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 11 | 12 | 12 | 12
Participants
  All reactogenicity: None | 10 | 6 | 9 | 8
  All reactogenicity: Mild | 1 | 5 | 3 | 4
  All reactogenicity: Moderate | 0 | 1 | 0 | 0
  Local reactogenicity: None | 11 | 7 | 9 | 8
  Local reactogenicity: Mild | 0 | 4 | 3 | 4
  Local reactogenicity: Moderate | 0 | 1 | 0 | 0
  Systemic reactogenicity: None | 10 | 9 | 12 | 11
  Systemic reactogenicity: Mild | 1 | 3 | 0 | 1
  Systemic reactogenicity: Moderate | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic or local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic); Test type: Equivalence — Equivalence defined as p<0.05; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.0000, Fisher Exact

5. Primary Outcome: Maximum Local or Systemic Reactogenicity After the Third Vaccination
Description: as for outcome 2
Time Frame: 7 days post Vaccination #3 on Day 56
Population: 44 subjects received third vaccination (4 less than Analysis Population Description). 2 subjects lost in Placebo group, one due to pain, swelling (after vaccination #2) and 1 due to incarceration. 1 subject lost from 10 μg cohort due to illness, 1 subject lost in 30 μg cohort because did not continue to meet inclusion/exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 10 | 11 | 11 | 12
Participants
  All reactogenicity: None | 9 | 7 | 9 | 8
  All reactogenicity: Mild | 1 | 3 | 2 | 3
  All reactogenicity: Moderate | 0 | 1 | 0 | 1
  Local reactogenicity: None | 10 | 8 | 10 | 8
  Local reactogenicity: Mild | 0 | 3 | 1 | 4
  Local reactogenicity: Moderate | 0 | 0 | 0 | 0
  Systemic reactogenicity: None | 9 | 8 | 9 | 9
  Systemic reactogenicity: Mild | 1 | 2 | 2 | 2
  Systemic reactogenicity: Moderate | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic or local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (systemic); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.0000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 10 μg P2-VP8 vs 30 μg P2-VP8 vs 60 μg P2-VP8; Proportion of subjects per Group with any Moderate or Higher Reaction (local reaction); Test type: Equivalence — Equivalence was defined as p<0.05; p = 1.0000, Fisher Exact

6. Secondary Outcome: Number and Percentage of Subjects With Anti-P2-VP8 Immunoglobulin G (IgG) and Immunoglobulin A (IgA) Seroresponses
Description: Seroresponse was defined as as a four-fold increase in antibody titers between baseline and 4-weeks post-third injection.
Time Frame: 4 weeks post 3rd immunization (84 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 11 | 12 | 12 | 12
Participants
  IgG: Seroresponse | 0 | 12 | 11 | 12
  IgG: No seroresponse | 11 | 0 | 1 | 0
  IgA: Seroresponse | 0 | 12 | 12 | 12
  IgA: No seroresponse | 11 | 0 | 0 | 0

7. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-P2-VP8 Immunoglobulin G (IgG)
Description: Measured from sera taken on Days 0, 28, 56 and 84 (before the first injection and 4 weeks after each injection).
Time Frame: Days 0, 28, 56 and 84 (before the first injection and 4 weeks after each injection)
Population: Included subjects that received vaccinations (see participant flow for reasons why some subjects did not receive all vaccinations).
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 12 | 12 | 12 | 12
titer
  Baseline | 519 [155 to 1740] | 362 [164 to 800] | 457 [270 to 773] | 285 [135 to 604]
  Pre-vaccination 2 | 551 [172 to 1761] | 2607 [1168 to 5821] | 4314 [2273 to 8190] | 2867 [1070 to 7686]
  Pre-vaccination 3: number analyzed (Participants) | 11 | 11 | 12 | 12
  Pre-vaccination 3 | 513 [140 to 1883] | 7373 [3470 to 15666] | 8489 [4670 to 15431] | 12438 [6365 to 24307]
  4 weeks post-vaccination 3: number analyzed (Participants) | 11 | 12 | 12 | 12
  4 weeks post-vaccination 3 | 520 [145 to 1870] | 13090 [5881 to 29135] | 13932 [7163 to 27097] | 19546 [10231 to 37343]

8. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-P2-VP8 Immunoglobulin A (IgA)
Description: Measured from sera taken on Days 0, 28, 56 and 84 (before the first injection and 4 weeks after each injection).
Time Frame: Days 0, 28, 56 and 84 (before the first injection and 4 weeks after each injection)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 12 | 12 | 12 | 12
titer
  Baseline | 519 [115 to 1740] | 362 [164 to 800] | 457 [270 to 773] | 285 [135 to 604]
  Pre-vaccination 2 | 551 [172 to 1761] | 2607 [1168 to 5821] | 4314 [2273 to 8190] | 2867 [1070 to 7686]
  Pre-vaccination 3: number analyzed (Participants) | 11 | 11 | 12 | 12
  Pre-vaccination 3 | 513 [140 to 1883] | 7373 [3470 to 15666] | 8489 [4670 to 15431] | 12438 [6365 to 24307]
  4 weeks post-vaccination 3: number analyzed (Participants) | 11 | 12 | 12 | 12
  4 weeks post-vaccination 3 | 520 [145 to 1870] | 13090 [5881 to 29135] | 13932 [7163 to 27097] | 19546 [10231 to 37343]

9. Secondary Outcome: Number and Percentage of Subjects With Serum Neutralizing Antibody Seroresponse, by Rotavirus Strain
Description: as for outcome 6
Time Frame: 4 weeks post 3rd immunization (84 days)
Measure: Count of Participants; unit: Participants
Arm/Group | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8
Number analyzed (Participants) | 12 | 12 | 12
Participants
  WA: Seroresponse | 8 | 5 | 7
  WA: No seroresponse | 4 | 7 | 5
  89-12: Seroresponse | 10 | 8 | 10
  89-12: No seroresponse | 2 | 4 | 2
  DS1: Seroresponse | 0 | 6 | 7
  DS1: No seroresponse | 12 | 6 | 5
  P: Seroresponse | 7 | 8 | 10
  P: No seroresponse | 5 | 4 | 2
  ST3: Seroresponse | 0 | 1 | 2
  ST3: No seroresponse | 12 | 11 | 10
  BRB: Seroresponse | 0 | 3 | 4
  BRB: No seroresponse | 12 | 9 | 8
  SC2: Seroresponse | 1 | 4 | 4
  SC2: No seroresponse | 11 | 8 | 8
  W161: Seroresponse | 8 | 9 | 10
  W161: No seroresponse | 4 | 3 | 2

ADVERSE EVENTS:
Time Frame: 6 months after final vaccination (224 days)
Arm/Group | 10 μg P2-VP8 | 30 μg P2-VP8 | 60 μg P2-VP8 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/12 | 5/12 | 7/12 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 μg P2-VP8 (N=12) | 30 μg P2-VP8 (N=12) | 60 μg P2-VP8 (N=12) | Placebo (N=12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 μg P2-VP8 (N=12) | 30 μg P2-VP8 (N=12) | 60 μg P2-VP8 (N=12) | Placebo (N=12)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 0 | 4
Vaginitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 3 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 2 | 1 | 1 | 1
White blood cell count increased (Investigations) | 1 | 2 | 0 | 3
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No